CLINICAL TRIAL: NCT05938621
Title: Estamos Juntos (We Are Together): Improving HIV Care Delivery by Capacitating Health Care Providers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Carolyn Audet, Associate Professor of Health Policy, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R34MH127975 (NIH)
Record Dates: First submitted 2023-06-28; First posted 2023-07-10 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Behavior Therapy; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard of Care (No Intervention): Health care providers in this arm will receive no intervention
- Resilience intervention (Experimental): Providers in this arm will receive training to improve their resilience and well-being
  Interventions: Behavioral: behavioral therapy and education
- Resilience and Stigma group (Experimental): Providers in this group will receive training to improve their resilience and well-being as well as receive sessions about the impact of stigmatizing their patients.
  Interventions: Behavioral: behavioral therapy and education
- Anti-stigma group (Experimental): Providers in this group will receive sessions focusing on the impact that stigmatizing patients can have on themselves and their patients. Strategies to minimize negative feelings will be developed.
  Interventions: Behavioral: behavioral therapy and education

INTERVENTIONS:
Behavioral: behavioral therapy and education — Sessions that focus on developing self-awareness and strategies to improve well-being will be the focus of the interventions.
  Arms: Anti-stigma group; Resilience and Stigma group; Resilience intervention

SUMMARY:
Health care workers' negative behavior towards patients (likely a reflection of low job satisfaction, frustration with delivering HIV care and treatment in extremely resource-limited settings, and burnout) is one of the primary reasons people living with HIV abandon treatment in Mozambique. The purpose of this proposal is to test the impact and implementation of a provider resilience intervention and an anti-stigma intervention, individually and in combination, using a randomized controlled trial design at four health facilities. This potentially high-impact intervention offers the opportunity to test a low-cost, provider-focused approach to improving HIV treatment that, if proven effective at increasing adherence and retention in care, could be tested in a fully powered R01 trial in Mozambique.

DETAILED DESCRIPTION:
Mozambique has made progress towards their 95-95-95 goals, yet only 65% of people newly initiated in HIV treatment remain in care at 12 months. HIV treatment adherence has been undermined by a lack of compassionate health care service delivery. People living with HIV in our study region of Zambezia province report being treated disrespectfully by health care workers as one of the leading causes of treatment abandonment. Common complaints include insulting patients' intellectual capacity, ignoring concerns with side effects or co-occurring infections, and refusing to treat patients seen as "unworthy". While health care worker behavior is appalling, it is likely a reflection of high rates of burnout, job dissatisfaction, and frustration with patients they perceive to be uncooperative.

The implementation of Estamos Juntos (We are Together) will allow us to test a multiprong intervention designed to address provider-barriers to delivering compassionate care via two synergistic components: (1) Resilience and well-being training for health care providers who have expressed low job satisfaction, frustration with delivering care in an extremely resource-limited setting, and burnout; and (2) Anti-stigma training for health care providers who see those with low socioeconomic status, low levels of education, and those living with HIV as "lesser-than" themselves. We propose to pilot test the implementation and impact of each psychosocial intervention individually, and in combination, using a randomized controlled trial design at four health facilities. We hypothesize that the facility where health care workers receive both resilience and anti-stigma training will see the greatest change in health care worker outcomes, including decreased stigmatizing attitudes, emotional exhaustion, and depersonalize of their patients, as well as increased resilience and job satisfaction. Patients receiving care and treatment from intervention providers will show increased retention and medication adherence, as well as improvements in health care services satisfaction, medical mistrust, and perceived stigma from health care providers.

ELIGIBILITY:
Provider Criteria

Inclusion Criteria:

* Adult individuals, 18 years of age or older;
* working as physicians, nurses, medical technicians, health counselors, community health care workers, or other clinical and non-clinical staff (e.g., receptionists, data entry clerk) who provide health services to adults living with HIV at one of the four study sites;
* willing to be followed as a study participant during the 6-month study period, and does not intend to transfer to another health facility (HF) during the study period (per investigator's assessment at time of recruitment), as self-reported.
* Be able to read and write in Portuguese, as self-reported.

Exclusion Criteria:

* Those who are not permanent members of the health facility staff (i.e., floating providers that work at multiple sites in a given week);
* Any clinical or mental condition, including the influence of drugs or alcohol at the time of study recruitment, that as per the investigator's opinion/assessment, would preclude the provision of informed consent or make study participation unsafe or unethical;
* Individuals working in the health facility but from the following cadres: drivers, security personnel, and workers with no patient-facing roles.

Patient Criteria

Inclusion:

* Adult individuals, 18 years of age or older
* Active in care (i.e., not in default)
* Receiving HIV care and treatment at one of the four study sites.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28448 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-02-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ministry of Health, Quelimane, Zambezia Province, Mozambique

IPD SHARING:
Plan to Share IPD: Undecided
Mozambique is in the process of determining what IPD can be shared to researchers not on the approved study team. Once we know their new legal process we will update this plan.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited 25 health care workers from each of four health facilities. Health care workers consented to participate and interacted with the study team. All eligible patients who they treated during the subsequent 6 months were included in the clinical outcome data.
Units Other Than Participants: Clinics
Period: Overall Study
Arm/Group | Standard of Care | Resilience Intervention | Resilience and Stigma Group | Anti-stigma Group
Started (Provider enrollment) | 25; 1 Clinics (In this site the 25 providers treated 4,597 patients) | 25; 1 Clinics (In this site, the 25 providers treated 12,904 patients) | 25; 1 Clinics (In this site, the 25 providers treated 6,324 patients) | 25; 1 Clinics (In this site, the 25 providers treated 4523 patients.)
Number of Patients Receiving Care | 4597; 1 Clinics | 12904; 1 Clinics | 6324; 1 Clinics | 4523; 1 Clinics
Completed (This is only information about the providers given that they were the ones who were formally enrolled in the trial) | 24; 1 Clinics (Only the providers are included in the number of people who completed the intervention.) | 20; 1 Clinics (Only the providers are included in the number of people who completed the intervention.) | 23; 1 Clinics (Only the providers are included in the number of people who completed the intervention.) | 23; 1 Clinics (Only the providers are included in the number of people who completed the intervention.)
Not Completed | 1; 0 Clinics | 5; 0 Clinics | 2; 0 Clinics | 2; 0 Clinics
Not completed — Lost to Follow-up | 1 | 5 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Provider Baseline Data and Patient Data are collapsed together here.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Resilience Intervention | Resilience and Stigma Group | Anti-stigma Group | Total
Number analyzed (Participants) | 4622 | 12929 | 6349 | 4548 | 28448
Age, Continuous [Mean (Standard Deviation); unit: years] — Provider Baseline Data Population: These data are from the 100 providers that were enrolled in the study
  years
    number analyzed (Participants) | 25 | 25 | 25 | 25 | 100
    (all) | 33.5 (7.09) | 33.8 (8.88) | 35.2 (8.18) | 33.7 (6.67) | 34.1 (7.67)
Age, Continuous [Mean (Standard Deviation); unit: years] — Patient Data Population: This is the data from patients only.
  years
    number analyzed (Participants) | 4597 | 12904 | 6324 | 4523 | 28348
    (all) | 32.3 (10.60) | 29.7 (18.86) | 32.11 (10.49) | 30.6 (10.11) | 30.8 (14.91)
Sex: Female, Male [Count of Participants; unit: Participants] — Provider Baseline Data Population: These data are from the 100 health care providers enrolled in the study
  Participants
    number analyzed (Participants) | 25 | 25 | 25 | 25 | 100
    Female | 16 | 13 | 19 | 15 | 63
    Male | 9 | 12 | 6 | 10 | 37
Sex: Female, Male [Count of Participants; unit: Participants] — These are data from the patients treated at the study sites Population: These data only include patients seen at the study clinics
  Participants
    number analyzed (Participants) | 4597 | 12904 | 6324 | 4523 | 28348
    Female | 3044 | 9058 | 4379 | 2926 | 19407
    Male | 1553 | 3846 | 1945 | 1597 | 8941
Race (NIH/OMB) [Count of Participants; unit: Participants] — Provider and Patient Baseline Data
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 4622 | 12929 | 6349 | 4548 | 28448
    White | 0 | 0 | 0 | 0 | 0
    More than one race | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Provider and Patient Baseline Data
  participants
    Mozambique | 4622 | 12929 | 6349 | 4548 | 28448
Number of Years Working in this Health Facility [Mean (Standard Deviation); unit: years] — Provider Baseline Data Population: This only includes provider data
  years
    number analyzed (Participants) | 25 | 25 | 25 | 25 | 100
    (all) | 3.4 (1.95) | 6.1 (6.05) | 5.5 (3.70) | 4.2 (3.09) | 4.8 (4.07)

OUTCOME MEASURES:

1. Primary Outcome: Burnout
Description: We assessed burnout using the Copenhagen Burnout Inventory (CBI) at baseline and again at 6 months. Higher numbers indicate greater levels of burnout. We are reporting the change in burnout scores from baseline to 6 months post-intervention. The scores can range from a minimum of 0 to a maximum of 100. We are reporting changes in scores, so some numbers are negative.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard of Care | Resilience Intervention | Resilience and Stigma Group | Anti-stigma Group
Number analyzed (Participants) | 24 | 20 | 23 | 23
units on a scale | -2.0 [-10.9 to 9.5] | -5.9 [-8.2 to -2.0] | -5.3 [-13.8 to 2.0] | -3.9 [-13.8 to 2.0]

ADVERSE EVENTS:
Time Frame: The data were collected from providers over a six-month period. Per protocol, adverse event data were not collected from patients.
Arm/Group | Standard of Care | Resilience Intervention | Resilience and Stigma Group | Anti-stigma Group
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-09-27): https://cdn.clinicaltrials.gov/large-docs/21/NCT05938621/Prot_SAP_ICF_001.pdf